CLINICAL TRIAL: NCT02548234
Title: Effect of Mirror Therapy Versus Bilateral Arm Training for Rehabilitation After Chronic Stroke: a Pilot Randomized-controlled Trial
Brief Title: Effect of Mirror Therapy Versus Bilateral Arm Training for Rehabilitation After Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH104-REC3-052
Record Dates: First submitted 2015-09-09; First posted 2015-09-14 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Stroke
Keywords: Stroke; Randomized control trial; Mirror therapy; Bilateral arm training; Comparative efficacy research; Neurorehabilitation
MeSH Terms: conditions — Stroke | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirror therapy (Experimental): Mirror therapy group received training for 1.5 hours/day, 3 days/week, for 4 weeks and home programs for 30-40 min/day, 5 days/week.
  Interventions: Other: Mirror therapy
- Bilateral arm training (Experimental): Bilateral arm training group received training for 1.5 hours/day, 3 days/week, for 4 weeks and home programs for 30-40 min/day, 5 days/week.
  Interventions: Other: Bilateral arm training

INTERVENTIONS:
Other: Mirror therapy — Mirror therapy group received training for 1.5 hours/day, 3 days/week, for 4 weeks and home programs for 30-40 min/day, 5 days/week.
  Arms: Mirror therapy
Other: Bilateral arm training — Bilateral arm training group received training for 1.5 hours/day, 3 days/week, for 4 weeks and home programs for 30-40 min/day, 5 days/week.
  Arms: Bilateral arm training

SUMMARY:
The study purpose is to compare the efficacy of mirror therapy and bilateral arm training on movement strategies of the affected upper extremity and functional outcome in chronic stroke patients.

DETAILED DESCRIPTION:
Study background: Approximately 80% of stroke survivors have an upper and/or lower limb impairment (Barker 1997), and impairment of the arm explains up to 50% of the variance in functional limitation after stroke. Brain imaging research using magnetoencephalography found that mirror therapy combined with bilateral arm training could potentially aid stroke rehabilitation by normalizing an asymmetrical pattern of movement-related beta desynchronization in primary motor cortex. However, different neural mechanisms may cause different effect of motor control recovery after the two different approaches, which have yet to be studied. Study purpose：To compare the efficacy of mirror therapy and bilateral arm training on movement strategies of the affected upper extremity and functional outcome in chronic stroke patients. Study method: This was a single-blind, randomized, comparative efficacy research. Sixty participants with chronic stroke will be recruited in the occupational therapy clinics at four hospitals and randomly assigned to the mirror therapy and bilateral arm training groups. The intervention will consist of 1.5 hrs/day, 5 days/wk for 4 wks, including 3 days of hospital-based therapy and 5 days of home practice. Primary outcomes were muscular properties (grip strength) and sensorimotor measurements. Secondary outcomes included measures of daily functions to gain insight about movement capabilities. The validity and reliability of all measurements have been proposed. Finally, the Mann-Whitney U test and the Fisher exact test will be used to compare the significant differences between the two approaches. The effect size of dependent variables will be reported also.

ELIGIBILITY:
Inclusion Criteria:

* more than 6 months after onset of an ischemic or hemorrhage stroke
* no excessive spasticity on all joints of the affected arm

Exclusion Criteria:

* history of stroke or other neurologic, neuromuscular, or orthopedic disease
* participation in other experimental rehabilitation or drug studies concurrent with this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-09-11 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

PRIMARY OUTCOMES:
The efficacy of mirror therapy versus bilateral arm training on sensorimotor functions | within four weeks (plus or minus 3 days) after intervention
  Revised Nottingham Sensory Assessment and Fugl-Meyer Assessment will be used to measure sensorimotor functions. The statistical analysis will be performed to compare the significant differences for the efficacy of mirror therapy versus bilateral arm training.

SECONDARY OUTCOMES:
The efficacy of mirror therapy versus bilateral arm training on motor performance | within four weeks (plus or minus 3 days) after intervention
  The Chedoke Arm and Hand Activity Inventory (CAHAI) will be used to measure arm and hand functions on real-life bilateral tasks. The statistical analysis will be performed to compare the significant differences for the efficacy of mirror therapy versus bilateral arm training on motor performance.
The efficacy of mirror therapy versus bilateral arm training on motor performance | within four weeks (plus or minus 3 days) after intervention
  Motor Activity Log (MAL) will be used to measure self-perceived real-world use. The statistical analysis will be performed to compare the significant differences for the efficacy of mirror therapy versus bilateral arm training.
The efficacy of mirror therapy versus bilateral arm training on quality of life | within four weeks (plus or minus 3 days) after intervention
  Stroke Impact Scale Version 3.0 (SIS) will be used to measure patient reported quality of life and multidimensional stroke recovery. The statistical analysis will be performed to compare the significant differences for the efficacy of mirror therapy versus bilateral arm training.

CONTACTS AND LOCATIONS:
Overall Officials: Keh-Chung Lin, ScD, Principal Investigator — National Taiwan University
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Thieme H, Mehrholz J, Pohl M, Behrens J, Dohle C. Mirror therapy for improving motor function after stroke. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD008449. doi: 10.1002/14651858.CD008449.pub2. PMID 22419334
- [Background] Wu CY, Huang PC, Chen YT, Lin KC, Yang HW. Effects of mirror therapy on motor and sensory recovery in chronic stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2013 Jun;94(6):1023-30. doi: 10.1016/j.apmr.2013.02.007. Epub 2013 Feb 15. PMID 23419791
- [Background] Samuelkamaleshkumar S, Reethajanetsureka S, Pauljebaraj P, Benshamir B, Padankatti SM, David JA. Mirror therapy enhances motor performance in the paretic upper limb after stroke: a pilot randomized controlled trial. Arch Phys Med Rehabil. 2014 Nov;95(11):2000-5. doi: 10.1016/j.apmr.2014.06.020. Epub 2014 Jul 23. PMID 25064777
- [Background] Wolf A, Scheiderer R, Napolitan N, Belden C, Shaub L, Whitford M. Efficacy and task structure of bimanual training post stroke: a systematic review. Top Stroke Rehabil. 2014 May-Jun;21(3):181-96. doi: 10.1310/tsr2103-181. PMID 24985386